CLINICAL TRIAL: NCT00909662
Title: Physiology of Chemotherapy Induced Fatigue and Cognitive Dysfunction in Early Stage Breast Cancer
Brief Title: Fatigue Caused by Chemotherapy in Women Who Have Undergone Surgery for Breast Cancer and in Healthy Volunteers
Status: Terminated | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE7107; P30CA043703 (NIH); CASE7107 (Other: Case Comprehensive Cancer Center); CASE-7107-CC400 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Fatigue; Long-term Effects Secondary to Cancer Therapy in Adults
Keywords: cognitive/functional effects; long-term effects secondary to cancer therapy in adults; fatigue; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Mental Status and Dementia Tests; Therapeutics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Female patients with operable breast cancer intending to undergo adjuvant chemotherapy
  Interventions: Procedure: assessment of therapy complications; Procedure: cognitive assessment; Procedure: fatigue assessment and management
- Participants: Female control subjects will be recruited, consisting predominantly of age-matched (i.e.+/- 10 years of age) friends or family members of the patients.
  Interventions: Procedure: assessment of therapy complications; Procedure: cognitive assessment; Procedure: fatigue assessment and management

INTERVENTIONS:
Procedure: assessment of therapy complications — 1. Questionnaires: Brief Fatigue Inventory, Brief Mental Fatigue and BDI FastScreen
  2. Cognitive Task (2 timed 2-minute tests) with Concomitant EEG
  3. Physical Task (Sustained Elbow Flexion) with Concomitant EEG and EMG plus TMS
  4. Borg 15-Category Scale
Procedure: cognitive assessment — Cognitive Task (2 timed 2-minute tests) with Concomitant EEG
Procedure: fatigue assessment and management — 1. Questionnaires: Brief Fatigue Inventory, Brief Mental Fatigue and BDI FastScreen
  2. Cognitive Task (2 timed 2-minute tests) with Concomitant EEG
  3. Physical Task (Sustained Elbow Flexion) with Concomitant EEG and EMG plus TMS
  4. Borg 15-Category Scale

SUMMARY:
RATIONALE: Gathering information over time from women undergoing chemotherapy for breast cancer may help doctors learn more about mental and physical fatigue caused by treatment.

PURPOSE: This clinical trial is studying fatigue caused by chemotherapy in women who have undergone surgery for stage I, stage II, or stage III breast cancer and in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess treatment-related fatigue, cognitive dysfunction, and recovery in women undergoing adjuvant chemotherapy for stage I-III breast cancer as compared with a patient-selected control population.
* To determine whether fatigue induced by sustained isometric contraction (SIC) is more of central or peripheral (muscular) origin in patients with and without treatment-related fatigue.
* To characterize changes from baseline in potential abnormal signal processing in the brain while performing cognitive-assessment testing (CAT) in patients experiencing chemotherapy-related cognitive dysfunction compared with the controls.

OUTLINE: Patients and participants undergo assessment of treatment-related fatigue and cognitive dysfunction (i.e., mental fatigue) at baseline, after completion of 3-4 courses of standard adjuvant chemotherapy, and 1-3 weeks after completion of the most recent treatment. Patient recovery will be assessed at approximately 1 year from baseline. Study assessments will include a brief fatigue inventory, a cognitive assessment, and muscle fatigability testing through a sustained isometric contraction. Additional assessments will include quantification of brain and muscle signal alterations in patients with and without treatment-related fatigue and cognitive-assessment testing in patients experiencing chemotherapy-related cognitive dysfunction.

Patients and participants also undergo collection of data to obtain information on patient age, body mass index, and menopausal status at baseline and at 1 year. Additional information is collected on type of chemotherapy treatment and any hormonal or other anticancer treatments administered throughout the course of the study. Cancer recurrences or new cancer events are also recorded.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets either of the following criteria:

  * Has completed surgery for stage I-III breast cancer AND meets the following criteria:

    * No bilateral axillary dissection
    * Clinically free of active disease
    * Planning to receive adjuvant chemotherapy for operable breast cancer
  * Friend or relative of patient matched for age (± 10 years) (control)
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Known menopausal status
* Able to read English
* No history of significant cardiovascular disease or stroke, polyneuropathy, amyotrophy, myosthenic syndrome, or pulmonary compromise
* Prior depression allowed provided that it was not significant
* Willing to come to the Cleveland Clinic for 3 assessments

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with operable breast cancer intending to undergo adjuvant chemotherapy will be enrolled from the outpatient oncology clinics of the Case Comprehensive Cancer Center.
  Twenty female control subjects will be recruited, consisting predominantly of age-matched (i.e.
  +/- 10 years of age) friends or family members of the patients.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Treatment-related fatigue as assessed by a brief fatigue inventory, a Brief Mental Fatigue Questionnaire, and a motor fatigability task with concurrent physiological measurements at baseline, during treatment, and 1 year after treatment completion | at baseline, after completion of 3-4 courses of standard adjuvant chemotherapy, and 1-3 weeks after completion of the most recent treatment.
Cognitive function as assessed by the Wechsler Adult Intelligence Scale III at baseline, during treatment, and 1 year after treatment completion | at baseline, after completion of 3-4 courses of standard adjuvant chemotherapy, and 1-3 weeks after completion of the most recent treatment.
Recovery at 1 year | at 1 year
Quantification of brain and muscle signal alteration in patients and controls with and without treatment-related fatigue as assessed by high-density EEG or EMG and force | measurements at baseline, during treatment, and 1 year after treatment completion
Characterization of potential abnormal signal processing in the brain in patients experiencing chemotherapy-related cognitive dysfunction as evaluated by cognitive-assessment testing and high-density EEG | measurements at baseline, during treatment, and 1 year after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Halle Moore, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Joseph Baar, MD, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio